CLINICAL TRIAL: NCT06515769
Title: Use of Thermography for the Prevention and Diagnosis of Rheumatic Foot
Acronym: TG-AR
Status: Not yet recruiting | Type: Observational
Sponsor: University of Seville (Other)
Responsible Party: Principal Investigator, ANA MARIA RAYO PEREZ, Principal Investigator, University of Seville
Other Study IDs: TERMOGRAPHYAR
Record Dates: First submitted 2024-06-24; First posted 2024-07-23 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Rheumatoid Arthritis; Rheumatoid Arthritis RA; Rheumatic Diseases
Keywords: Rheumatic foot; Rheumatoid Arthritis; Rheumatic diseases; Thermoghrapy
MeSH Terms: conditions — Arthritis, Rheumatoid; Rheumatic Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control group: healthy subjects: Subjects without rheumatoid arthritis or symptoms compatible with this disease
  Interventions: Diagnostic Test: TERMOGRAPHY
- Case group: subjects with rheumatoid arthritis: Subjects diagnosed with rheumatoid arthritis
  Interventions: Diagnostic Test: TERMOGRAPHY

INTERVENTIONS:
Diagnostic Test: TERMOGRAPHY — Obtaining an image of the foot using a thermographic camera

SUMMARY:
The aim of this observational study is to establish normal thermographic parameters in patients with rheumatoid arthritis, in order to prevent and diagnose rheumatic foot using thermography. The main question to be answered is: What are the normal thermographic parameters in rheumatic foot?

If there is a comparison group: the researchers will compare the thermography of the foot in healthy subjects and in subjects with rheumatoid arthritis to see if there are any alterations in the thermographic image.

Patients who wish to participate in the study will undergo a thermographic study of the foot, which does not entail any risk to their health.

ELIGIBILITY:
Inclusion Criteria:

* Patients with rheumatoid arthritis of more than 5 years' duration
* Healthy patients without diagnosed systemic disease
* Patients between 40 and 80 years of age

Exclusion Criteria:

* Patients who are pregnant or may become pregnant
* Patients with degenerative diseases or significant cognitive impairment
* Patients with rheumatic diseases without a diagnosis of rheumatoid arthritis

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Selected patients will be healthy subjects and subjects with more than 5 years of rheumatoid arthritis who wish to voluntarily participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
NORMAL PARAMETERS IN THERMOGRAPHY IN PATIENS WITH HEALTHY FOOT | One measurement will be taken at the start of the study and another measurement the following 6 month.
  Normal parameters of the healthy foot in thermography

SECONDARY OUTCOMES:
NORMAL PARAMETERS IN TERMOGRAPHY IN PATIENS WITH RHEUMATIC FOOT | One measurement will be taken at the start of the study and another measurement the following 6 month
  Normal parameters in thermography in patients with rheumatic foot

CONTACTS AND LOCATIONS:
Locations (1):
- University of Seville, Seville, Spain

IPD SHARING:
Plan to Share IPD: No